CLINICAL TRIAL: NCT02989805
Title: Engaging Patients With Mental Disorders From the ED in Outpatient Care: A Comparative Effectiveness Workforce Study of Peer Specialist vs. Professional Care Managers
Brief Title: Engaging Patients With Mental Disorders From the ED in Outpatient Care
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Benjamin Druss, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00091841
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-02

CONDITIONS: Mental Disorder
Keywords: Emergency Medicine; Psychiatry; Health Promotion; Public Health
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Professional Care Manager (Active Comparator): Each participating site will have a nurse or social worker to provide care management. Training activities will include modules for each of the key domains covered in the intervention: shared decision making, action planning; motivational interviewing; and mental health as a cornerstone of recovery, working effectively within the mental health system; and self-care and stress management.
  Interventions: Behavioral: Care Management
- Peer Specialist Care Manager (Experimental): Each participating site will have a peer specialist to provide care management. Peer specialists will have a minimum of a high school education, a history of a mental illness, be self-described as 'in recovery,' and have reliable transportation to the study site. All certified peer specialists will receive training in a curriculum that supports identifying and pursuing goals for recovery; developing and documenting recovery-focused treatment plans; and supporting linkages with community-based services. Peers learn to help other individuals with mental health conditions to facilitate mental health dialogues; explore mental health choices and options; identify and work with a clinician; and obtain access to community health supports.
  Interventions: Behavioral: Care Management

INTERVENTIONS:
Behavioral: Care Management — Professionals and peers will each deliver the same intervention. The intervention combines a traditional medical model of care management with a recovery-based approach.

SUMMARY:
This study will compare the effectiveness of professional and peer care managers in improving linkage to and engagement in outpatient care after an emergency department (ED) discharge, as well as the mechanisms by which engagement occurs. The study will use a multi-site randomized trial study design across 8 EDs in South Carolina with telepsychiatry programs; each site will have one professional care manager (social worker or nurse) and one peer specialist care manager. Eligible subjects at each site will be randomized to a one-year treatment engagement intervention, the Coordination, Access, Referral and Evaluation (CARE) Program with either a peer or professional care manager, resulting in a total of 290 participants across sites. The CARE program will focus on shared decision-making between care managers and patients, and combines the traditional medical model of care management with a recovery-based approach.

DETAILED DESCRIPTION:
Existing literature indicates that there is potential effectiveness of care management delivered by mental health professionals in improving treatment engagement and reducing inpatient readmissions and that certified peer specialists may be able to deliver an array of mental health services of similar or better quality as mental health professionals. However, there have been no studies comparing certified peer specialists to professionals in interventions to increase treatment engagement and reduce readmissions. This study will be the first to examine the potential benefits and tradeoffs between these two groups of providers.

There is an urgent need to improve care transitions for patients with mental disorders seen in emergency departments (ED). Care management can improve treatment engagement after ED discharge for patients with mental disorders, and certified peer specialists hold promise in providing these services. However, there are no data comparing care management delivered by peers and professionals in these settings. With funding from a Patient-Centered Outcomes Research Institute (PCORI) grant the study team will be able to implement a manualized care management program to improve follow-up and treatment engagement for patients in South Carolina, supported by preliminary data and experience from work previously conducted by the study team.

The overall goal of the project is to compare the effectiveness of professional and peer care managers in improving linkage to and engagement in outpatient care after an ED discharge, as well as the mechanisms by which engagement occurs. The study will use a multi-site randomized trial study design across 8 EDs in South Carolina with telepsychiatry programs; each site will have one professional care manager (social worker or nurse) and one peer specialist care manager. Eligible subjects at each site will be randomized to a one-year treatment engagement intervention, namely the Coordination, Access, Referral and Evaluation (CARE) Program with either a peer or professional care manager, resulting in a total of 290 participants. The CARE program will focus on shared decision-making between care managers and patients, and combines the traditional medical model of care management with a recovery-based approach.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the emergency department for a primary diagnosis of a mental disorder
* Plan for discharge to a participating community mental health center (CMHC)
* Lives within the CMHC catchment area

Exclusion Criteria:

* Cognitive impairment
* Not able to speak English
* Admission to the hospital from the emergency department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Druss, MD, Principal Investigator — Emory University
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began in April 2017 and all follow-up visits were complete by December 31, 2019. Participants were enrolled from the patient population at 8 emergency departments in South Carolina.
Groups:
- Professional Care Manager: Participants meeting with a nurse or social worker to provide care management
- Peer Specialist Care Manager: Participants meeting with a peer specialist to provide care management
Period: Overall Study
Arm/Group | Professional Care Manager | Peer Specialist Care Manager
Started | 160 | 166
Completed | 154 | 162
Not Completed | 6 | 4
Not completed — invalid consent | 6 | 4

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Professional Care Manager | Peer Specialist Care Manager | Total
Number analyzed (Participants) | 154 | 162 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (12.6) | 33.9 (10.2) | 35.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 85 | 170
  Male | 69 | 77 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 19
  Not Hispanic or Latino | 146 | 151 | 297
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 67 | 60 | 127
  White | 78 | 88 | 166
  More than one race | 6 | 10 | 16
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 154 | 162 | 316

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Attending at Least One Outpatient Visit
Description: This outcome was operationally measured as at least one outpatient visit for a mental health problem in the 30 days after discharge from the emergency department. Data were obtained from the South Carolina Office of Revenue and Fiscal Affairs (RFA). The RFA data warehouse pulls client-specific data from an array of health and human services facilities, agencies and organizations and makes possible the integration of data from disparate sources at the client level by means of an internally assigned unique tracking number.
Time Frame: 30 days after discharge
Population: Participants completing the study are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Professional Care Manager | Peer Specialist Care Manager
Number analyzed (Participants) | 154 | 162
Participants | 85 | 70

2. Secondary Outcome: Percentage of Outpatient Visits Attended
Description: Outpatient engagement will be assessed by the percentage of outpatient visits attended.
Time Frame: 6 months after discharge
Population: This analysis includes participants who had at least one visit scheduled.
Measure: Mean (Standard Deviation); unit: percentage of visits attended
Arm/Group | Professional Care Manager | Peer Specialist Care Manager
Number analyzed (Participants) | 94 | 92
percentage of visits attended | 66.9 (24.9) | 66.2 (27.9)

3. Secondary Outcome: Number of Participants Being Readmitted to the Emergency Room
Description: The number of emergency room readmissions, for mental health/substance use and all-cause emergency room visits, is presented here.
Time Frame: 6 months after discharge
Population: This analysis includes participants for whom the 6-month follow-up data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Professional Care Manager | Peer Specialist Care Manager
Number analyzed (Participants) | 131 | 134
Participants | 77 | 77

4. Secondary Outcome: Number of Participants Being Admitted for Inpatient Hospitalization
Description: The number of inpatient hospitalizations, for mental health problems as well as all cause patient admissions, is presented here.
Time Frame: 6 months after discharge
Population: This analysis includes participants for whom the 6-month follow-up data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Professional Care Manager | Peer Specialist Care Manager
Number analyzed (Participants) | 131 | 134
Participants | 28 | 35

ADVERSE EVENTS:
Time Frame: All-cause mortality events were collected from the time participants gave consent to take part in the study through the 6-month follow-up visit.
Description: Only data on all-cause mortality events were collected during this study. All mortality events were reported to the Data Safety and Monitoring Board (DSMB) for review.
Arm/Group | Professional Care Manager | Peer Specialist Care Manager
All-Cause Mortality (participants affected / at risk) | 3/154 | 2/162
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT02989805/Prot_SAP_ICF_000.pdf